CLINICAL TRIAL: NCT02608957
Title: Evaluation of the Latella™ Knee Implant System for Medial Osteoarthritis Pain Reduction (Latella-US Study)
Brief Title: Evaluation of the Latella™ Knee Implant System for Medial Osteoarthritis Pain Reduction
Acronym: Latella-US
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor elected to terminate the study prior to subject treatment.
Sponsor: Cotera, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP-0002
Record Dates: First submitted 2015-11-13; First posted 2015-11-20 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Latella Knee Implant System (Experimental)
  Interventions: Device: Latella Knee Implant System

INTERVENTIONS:
Device: Latella Knee Implant System

SUMMARY:
The objective of the Latella-US study is to demonstrate the safety and efficacy of the Latella Knee Implant System for the reduction of medial osteoarthritis pain.

ELIGIBILITY:
Inclusion Criteria:

* History of pain due to medial osteoarthritis
* Qualifying baseline pain scores
* Kellgren-Lawrence Grades 2-3

Exclusion Criteria:

* Osteoporosis
* Rheumatoid arthritis
* Joint instability
* Metal ion allergy
* Permanent implant in or around the knee joint
* Prior anterior cruciate ligament reconstruction

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Primary Efficacy Endpoint: Mean change in KOOS pain score at 6 months | 6 Months
  Mean change in KOOS pain score at 6 months after treatment with the Latella Implant.
Primary Safety Endpoint: Surgical re-intervention rate at 6 months | 6 Months
  Surgical re-intervention rate during the 6 month period following implantation of the Latella device.

SECONDARY OUTCOMES:
Change in KOOS function score | 6, 12 and 24 months
Change in medial knee pain NRS (while walking) | 6, 12 and 24 months
Change in IKDC score | 6, 12 and 24 months
Device-related complications rate | 24 months
KOOS responder rate based on OARSI-OMERACT criteria | 6, 12 and 24 months
Proportion of subjects reaching MCID in KOOS pain score | 6, 12 and 24 months
Change in KOOS pain score | 12 and 24 months
Surgical re-intervention rate | 12 and 24 months
Procedure-related complications rate | 24 Months

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - The George Washington University, Washington D.C., District of Columbia
  - Rush University Medical Center, Chicago, Illinois